CLINICAL TRIAL: NCT03842033
Title: Implementing a Guidelines-Based M-Health Intervention for High Risk Asthma Patients
Acronym: PEAKmAAP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 206110; 1R01NR015988-01A1 (NIH)
Record Dates: First submitted 2017-05-15; First posted 2019-02-15 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Pediatric Asthma
Keywords: Asthma Action Plan; Smartphone App

STUDY DESIGN:
Intervention Model Description: We will conduct a randomized, controlled trial of 372 adolescents with uncontrolled mild-severe persistent asthma to examine the effectiveness of a personalized, interactive PEAKmAAP application with and without PCP data sharing in reducing asthma morbidity. The trial includes 3 groups: 1) a group utilizing the PEAKmAAP alone, 2) a group utilizing the PEAKmAAP with PCP data sharing (PEAKmAAP-DS), and 3) a usual care NutriMapgroup utilizing an application with daily non-asthma related reminders for attention control.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PEAKmAAP (Other): The Pulmonary Education and Asthma Knowledge mobile asthma action plan (PEAKmAAP) group will use a mobile "app" that will help manage asthma. Participants will be asked to enter asthma symptoms or peak flow every day. The PEAKmAAP guides participants when to take asthma medicines and sends reminders to take their medicines every day. mAAP also provides reminders when to get asthma medicines refilled. Asthma education messages and video links are also pushed via notification.
  Interventions: Behavioral: PEAKmAAP
- PEAKmAAP-Data Sharing (DS) (Other): PEAKmAAP with Data Sharing (PEAKmAAP-DS) group will be asked to enter asthma symptoms or peak flow every day. The PEAKmAAP guides participants when to take asthma medicines and sends reminders to take their medicines every day. PEAKmAAP also provides reminders when to get asthma medicines refilled. Asthma education messages and video links are also pushed via notification. The primary care provided (PCP) will receive monthly reports to help them know how the participant's asthma symptoms are over time.
  Interventions: Behavioral: PEAKmAAP-DS
- Nutrition Map (NutriMap) Usual Care (Other): Participants in this arm will use a smartphone application that sends daily non-asthma-related reminder for attention control. Participants will be asked to log their daily fruits and vegetables eaten. Participants will answer survey questions about their asthma and symptoms management.
  Interventions: Behavioral: NutriMap Usual Care

INTERVENTIONS:
Behavioral: PEAKmAAP — The PEAKmAAP group will use a mobile "app" that will help manage asthma.
  Arms: PEAKmAAP
Behavioral: PEAKmAAP-DS — This group will use the mobile app to help manage asthma. the primary care provider will receive monthly reports to help him/her know how the participants asthma symptoms are over time.
  Arms: PEAKmAAP-Data Sharing (DS)
Behavioral: NutriMap Usual Care — This group will use a non-asthma related app daily to record their daily intake of fruits and vegetables.
  Arms: Nutrition Map (NutriMap) Usual Care

SUMMARY:
The goal of this research study is to test how good an app is in making asthma easier to manage for 372 adolescents/young adults. The app is a mobile version of the asthma action plan.

DETAILED DESCRIPTION:
The proposed project aligns with our prior work targeting high-risk pediatric asthma populations in non-inner city environments by targeting adolescents at risk for future exacerbations from the Patient-Centered Medical Home (PCMH) at Arkansas Children's Hospital (ACH).

We propose to conduct a 3-arm randomized, controlled trial with 372 adolescents with uncontrolled asthma to test the effectiveness of mAAP. mAAP provides real-time, personalized feedback, asthma education, and data logging/tracking capabilities.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥12 and <21 years
* Persistent asthma according to national guidelines criteria
* Asthma Control Test (ACT) score ≤19
* Prescribed a preventive (controller) asthma medication in the past 6 months
* Access to a smartphone compatible with the PEAKmAAP and NutriMap
* Access to the internet
* Able to read and speak English

Exclusion Criteria:

* Significant underlying respiratory disease other than asthma, such as cystic fibrosis
* Significant co-morbid conditions, such as moderate to severe developmental delay that could interfere with the adolescent's ability to self-monitor asthma
* Current smoker
* Participation in the investigator's or other asthma clinical trials in the previous 6 months

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 370 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Asthma Control Test (ACT) Score | 3 months
  The primary outcome measure will be the change from ACT score ≤19 (uncontrolled asthma) to ACT >19 (controlled asthma) at 3 months.
  ACT is a validated five question survey that computes a number indicating asthma control. The instrument range is 1-25, with 25 indication well controlled asthma. A score of less than or equal 19 is considered poorly controlled asthma.

SECONDARY OUTCOMES:
Mediators of Asthma Control | 12 months
  Medication adherence and asthma self-efficacy. Pharmacy profiles will be accessed to determine medication adherence. We plan to administer the Pediatric Quality of Life (PedsQOL) to determine asthma self-efficacy. We plan to evaluate if participants are more likely to receive step up therapy per the national asthma guidelines.
Healthcare Utilization | 12 months
  We plan to utilize the PedsQOL instrument to measure participant quality of life. The PedQOL is a modular approach to measuring health related quality of life in children and adolescents with acute chronic health conditions. The instrument has a disease specific module for asthma. The instrument access four scales: physical functioning, emotional functioning, social functioning and school functioning.
Change in Asthma Control Test (ACT) Score to Access Secondary Outcomes | 12 months
  ACT a validated five question survey that computes a number indicating asthma control. The instrument range is 1-25, with 25 indicating well controlled asthma. A score of less than or equal 19 is considered poorly controlled asthma. We plan to prospectively assess clinical outcomes including ACT score, Composite Asthma Severity Index (CASI) score, acute healthcare utilization, medication use, and lung function. ACT scores may improve but remain ≤19 for participants with very poorly controlled asthma, we will assess for change in ACT score that is considered to be clinically important (as indicated by ≥3 point increase).The ACT score will be assessed via mobile survey to measure for sustained improvement throughout the study. We hypothesize that PCP data sharing will facilitate asthma control by alerting the PCP when asthma is worsening or failing to improve. The impact of PCP data sharing on ACT score will be measured to assess whether data sharing has added benefit to PEAKmAAP alone.
Composite Asthma Severity Index (CASI) score | 12 months
  The CASI quantify disease severity by looking at impairment risk and the amount of medication needed to maintain control. The CASI includes the major domains of asthma namely, impairment, as measured by day and night symptoms, along with albuterol use; and risk measured by forced expiratory volume in one second (FEV1) percent predicted and past asthma exacerbations, both of which are important predictors of future exacerbations.
Asthma Control Classification | 12 months
  Asthma guidelines categorize asthma control for individuals ≥12 years into 3 categories: well-controlled (WC), not well-controlled (NWC), or very poorly controlled (VPC). Asthma control is defined by the degree to which asthma manifestations are minimized by therapeutic intervention. Components of asthma control include measures of daytime symptoms, nighttime awakenings, activity limits, rescue medication use, and exacerbations requiring oral systemic corticosteroids. An assessment of asthma control will be made during the eligibility screening, at the in-person, structured interviews at baseline, 3 months and 12 months as well as via mobile survey at 6 and 9 months for all participants.
Lung Function and Airway Inflammation | 12 months
  Spirometry is the test most used for the assessment of the risk for adverse events and impairment in asthma. Forced expiratory volume in the first second (FEV1) expressed as percent predictive of reference population value or as a proportion of the forced vital capacity (FEV1/FVC) will be assessed. FeNO is a quantitative, non-invasive measure of airway inflammation that predicts responsiveness and adherence to ICS. We will measure lung function and FeNO at baseline, 3 months, and 12 months for all participants.

CONTACTS AND LOCATIONS:
Overall Officials: Tamara T. Perry, MD, Principal Investigator — University of Arkansas
Locations (1):
- Arkansas Children's Hospital Research Institute, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] MacDonald P. Understanding and treating asthma in adolescents. Paediatr Nurs. 2003 Feb;15(1):34-6. No abstract available. PMID 12655953
- [Background] Naimi DR, Freedman TG, Ginsburg KR, Bogen D, Rand CS, Apter AJ. Adolescents and asthma: why bother with our meds? J Allergy Clin Immunol. 2009 Jun;123(6):1335-41. doi: 10.1016/j.jaci.2009.02.022. Epub 2009 Apr 22. PMID 19395075
- [Background] Braun-Fahrlander C, Gassner M, Grize L, Minder CE, Varonier HS, Vuille JC, Wuthrich B, Sennhauser FH. Comparison of responses to an asthma symptom questionnaire (ISAAC core questions) completed by adolescents and their parents. SCARPOL-Team. Swiss Study on Childhood Allergy and Respiratory Symptoms with respect to Air Pollution. Pediatr Pulmonol. 1998 Mar;25(3):159-66. doi: 10.1002/(sici)1099-0496(199803)25:33.0.co;2-h. PMID 9556007
- [Background] Venn A, Lewis S, Cooper M, Hill J, Britton J. Questionnaire study of effect of sex and age on the prevalence of wheeze and asthma in adolescence. BMJ. 1998 Jun 27;316(7149):1945-6. doi: 10.1136/bmj.316.7149.1945. No abstract available. PMID 9641931
- [Background] Forero R, Bauman A, Young L, Larkin P. Asthma prevalence and management in Australian adolescents: results from three community surveys. J Adolesc Health. 1992 Dec;13(8):707-12. doi: 10.1016/1054-139x(92)90068-m. PMID 1290773
- [Background] Kyngas HA. Compliance of adolescents with asthma. Nurs Health Sci. 1999 Sep;1(3):195-202. doi: 10.1046/j.1442-2018.1999.00025.x. PMID 10894643
- [Background] Raherison C, Tunon-de-Lara JM, Vernejoux JM, Taytard A. Practical evaluation of asthma exacerbation self-management in children and adolescents. Respir Med. 2000 Nov;94(11):1047-52. doi: 10.1053/rmed.2000.0888. PMID 11127490
- [Background] Buston KM, Wood SF. Non-compliance amongst adolescents with asthma: listening to what they tell us about self-management. Fam Pract. 2000 Apr;17(2):134-8. doi: 10.1093/fampra/17.2.134. PMID 10758075
- [Background] Blaakman SW, Cohen A, Fagnano M, Halterman JS. Asthma medication adherence among urban teens: a qualitative analysis of barriers, facilitators and experiences with school-based care. J Asthma. 2014 Jun;51(5):522-9. doi: 10.3109/02770903.2014.885041. Epub 2014 Feb 7. PMID 24494626
- [Background] McQuaid EL, Kopel SJ, Klein RB, Fritz GK. Medication adherence in pediatric asthma: reasoning, responsibility, and behavior. J Pediatr Psychol. 2003 Jul-Aug;28(5):323-33. doi: 10.1093/jpepsy/jsg022. PMID 12808009
- [Background] Moorman JE, Rudd RA, Johnson CA, King M, Minor P, Bailey C, Scalia MR, Akinbami LJ; Centers for Disease Control and Prevention (CDC). National surveillance for asthma--United States, 1980-2004. MMWR Surveill Summ. 2007 Oct 19;56(8):1-54. PMID 17947969
- [Derived] Perry TT, Turner JH, Berlinski A, Simmons LA, Brown RH, Neal K, Marshall SA, He X, Chung S, Brown A, Spencer Rd HJ, Bian J. Comparing a Guideline-Based Mobile Health Intervention Versus Usual Care for High-Risk Adolescents With Asthma: Protocol of a Randomized Controlled Trial. JMIR Res Protoc. 2025 Jul 25;14:e69903. doi: 10.2196/69903. PMID 40712131